CLINICAL TRIAL: NCT00968981
Title: A Phase Ib, Open-Label, Dose-Scheduling Study of Hedgehog Pathway Inhibitor GDC-0449 in Patients With Locally Advanced or Metastatic Solid Tumors That Are Refractory to Standard Therapy or for Whom No Standard Therapy Exists
Brief Title: A Study of Hedgehog Pathway Inhibitor GDC-0449 in Patients With Locally Advanced or Metastatic Solid Tumors That Are Refractory to Standard Therapy or for Whom No Standard Therapy Exists
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHH4610g
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Solid Cancers
Keywords: Hedgehog; BCC; basal cell carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

ARMS (3):
- A (Experimental)
  Interventions: Drug: GDC-0449
- B (Experimental)
  Interventions: Drug: GDC-0449
- C (Experimental)
  Interventions: Drug: GDC-0449

INTERVENTIONS:
Drug: GDC-0449 — Daily oral repeating dose
  Arms: A
Drug: GDC-0449 — Three times weekly oral repeating dose
  Arms: B
Drug: GDC-0449 — Once weekly oral repeating dose
  Arms: C

SUMMARY:
This is a two stage, Phase Ib study designed to describe the pharmacokinetics of GDC-0449 in patients with advanced solid tumors that are refractory to treatment or for whom no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria

* Histologically documented, incurable, locally advanced or metastatic solid malignancy that has progressed after first-line and second-line therapy (if there is a second-line therapy that has been shown to provide clinical benefit); patients with basal cell carcinoma will be excluded from this study unless they do not qualify for another open GDC-0449 clinical trial
* For patients with disease that is evaluable by physical examination only, diagnosis must also include biomarker confirmation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Documented negative pregnancy test for women of childbearing potential and agreement to use an effective form of contraception for the duration of the study
* Adequate hematopoietic capacity
* Adequate hepatic function
* Adequate renal function
* At least 3 weeks since last chemotherapy, investigational agent, radiation therapy, or major surgical procedure and recovery to pre-treatment baseline or stabilization of all treatment-related toxicities

Exclusion Criteria

* Known, untreated central nervous system (CNS) malignancies or treated brain metastases that are not radiographically stable for ≥ 3 months
* Active infection requiring intravenous (IV) antibiotics
* Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, or current known active infection with hepatitis
* Any medical condition or diagnosis that would likely impair absorption of an orally administered drug (e.g., gastrectomy, ileal bypass, chronic diarrhea, gastroparesis)
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications
* Pregnant or lactating
* Treatment with excluded medications, including strong CYP450 inhibitors and inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Low, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Jia G, Chandriani S, Abbas AR, DePianto DJ, N'Diaye EN, Yaylaoglu MB, Moore HM, Peng I, DeVoss J, Collard HR, Wolters PJ, Egen JG, Arron JR. CXCL14 is a candidate biomarker for Hedgehog signalling in idiopathic pulmonary fibrosis. Thorax. 2017 Sep;72(9):780-787. doi: 10.1136/thoraxjnl-2015-207682. Epub 2017 Mar 1. PMID 28250200

RESULTS

PARTICIPANT FLOW:
Groups:
- GDC-0449 150 mg QD: Single dose of GDC-0449 150 mg capsule orally on Day 1 and then one capsule once daily (QD) orally from Day 4 to Day 14 (loading dose) followed by 150 mg capsule QD orally from Day 15 to Day 57 (maintenance dose).
- GDC-0449 150 mg TIW: Single dose of GDC-0449 150 mg capsule orally on Day 1 and then one capsule three times weekly (TIW) orally from Day 4 to Day 14 (loading dose) followed by 150 mg capsule TIW orally from Day 15 to Day 57 (maintenance dose).
- GDC-0449 150 mg QW: Single dose of GDC-0449 150 mg capsule orally on Day 1 and then one capsule once weekly (QW) orally from Day 4 to Day 14 (loading dose) followed by 150 mg capsule QW orally from Day 15 to Day 57 (maintenance dose).
Period: Overall Study
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Started | 23 | 22 | 22
Pharmacokinetic(PK) Evaluable Population | 20 (Participants with sufficient data to ensure reliable estimation of PK for at least Day 1 PK profile.) | 21 (Participants with sufficient data to ensure reliable estimation of PK for at least Day 1 PK profile.) | 22 (Participants with sufficient data to ensure reliable estimation of PK for at least Day 1 PK profile.)
Completed | 1 | 0 | 0
Not Completed | 22 | 22 | 22
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Disease Progression | 14 | 16 | 13
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 5 | 3 | 5
Not completed — Withdrawal by Subject | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants were included for baseline parameters.
Groups:
- GDC-0449 150 mg QD: Single dose of GDC-0449 150 mg capsule orally on Day 1 and then one capsule QD orally from Day 4 to Day 14 (loading dose) followed by 150 mg capsule QD orally from Day 15 to Day 57 (maintenance dose).
- GDC-0449 150 mg TIW: Single dose of GDC-0449 150 mg capsule orally on Day 1 and then one capsule TIW orally from Day 4 to Day 14 (loading dose) followed by 150 mg capsule TIW orally from Day 15 to Day 57 (maintenance dose).
- GDC-0449 150 mg QW: Single dose of GDC-0449 150 mg capsule orally on Day 1 and then one capsule QW orally from Day 4 to Day 14 (loading dose) followed by 150 mg capsule QW orally from Day 15 to Day 57 (maintenance dose).
- Total: Total of all reporting groups
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW | Total
Number analyzed (Participants) | 23 | 22 | 22 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.4) | 64.0 (12.3) | 62.9 (10.3) | 63.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 10 | 29
  Male | 13 | 13 | 12 | 38

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Disease Progression or Death
Description: Disease progression (assessed by Response Evaluation Criteria in Solid Tumors [RECIST]) was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions or the appearance of one or more new lesions and/or unequivocal progression of existing non target lesions.
Time Frame: Screening, Day 57, and every 8 weeks thereafter up to 52 weeks
Population: Efficacy Evaluable Population: all participants who had measurable disease at baseline and either had at least one follow-up tumor assessment or discontinued the study due to disease progression.
Measure: Number; unit: percentage of participants
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Number analyzed (Participants) | 17 | 20 | 20
percentage of participants | 52.9 | 75.0 | 40.0

2. Secondary Outcome: Percentage of Participants With a Response by Best Overall Response (BOR)
Description: BOR was defined as the best overall response observed during the treatment period according to RECIST. CR: disappearance of all TLs, with any pathological lymph nodes (whether target or non-target) having a reduction in short axis to less than 10 mm. PR: at least a 30% decrease in the sum of diameters of TLs, taking as reference the BL sum diameters. Progressive disease (PD): at least a 20% increase in the sum of diameters of TLs, taking as a reference the smallest sum on study (this included the baseline sum if that is the smallest on study). In addition to the relative increase in 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Stable disease (SD) was defined as neither sufficient shrinkages to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Screening Day 57, and every 8 weeks thereafter up to 52 weeks
Population: Efficacy Evaluable Population; only participants with measurable disease at baseline were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Number analyzed (Participants) | 13 | 18 | 15
percentage of participants
  Complete Response | 0.0 | 0.0 | 0.0
  Partial Response | 7.7 | 0.0 | 0.0
  Stable Disease | 30.8 | 22.2 | 53.3
  Progressive Disease | 61.5 | 77.8 | 40.0
  Unevaluable (UE) | 0.0 | 0.0 | 6.7

3. Secondary Outcome: Progression-Free Survival (PFS) Time
Description: PFS defined as the time from study treatment initiation to the first occurrence of disease progression, as determined by the investigator review of tumor assessments using RECIST, or death from any cause during the study (i.e., within 30 days after the last dose of study treatment).
Time Frame: Screening Day 57, and every 8 weeks thereafter up to 52 weeks
Population: Efficacy Evaluable Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Number analyzed (Participants) | 17 | 20 | 20
months | 1.9 [1.45 to 2.04] | 1.9 [1.84 to 1.97] | 2.2 [1.74 to 4.01]

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) at Steady-State for Both Total and Unbound GDC-0449
Time Frame: Predose and 1, 2, 4, 6, 24, 48, and 72 on Days 1, 29, 50, and 54 and predose on Days 8, 10, 15, 22, 33, 36, 43, and 57
Population: The PK Evaluable Population. Number of participants analyzed (N) is equal to (=) participants with baseline and at least one post-baseline assessment for this outcome; n = participants evaluable at specified time-points.
Measure: Median (Full Range); unit: hours
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Number analyzed (Participants) | 15 | 18 | 18
hours
  Total: Days 29-36 (n=15,18,18) | 24 [1 to 168] | 72 [0 to 96] | 15 [1 to 96]
  Total: Days 50-57 (n=11,13,10) | 74 [4 to 164] | 74 [4 to 164] | 24 [4 to 74]
  Unbound; Days 29-36 (n=15, 18, 18) | 24 [0 to 168] | 6 [0 to 168] | 6 [1 to 72]
  Unbound: Days 50-57 (n=11,13,10) | 104 [4 to 164] | 94 [4 to 104] | 4 [4 to 74]

5. Primary Outcome: Number of Participants With Greater Than (>) 50 Percent (%) Decrease in Trough Concentration at Steady State (Css, Trough)
Description: Percent change = ([trough concentration on Day 15 minus trough concentration on Day 57] divided by trough concentration on Day 15) multiplied by 100.
Time Frame: Predose and 1, 2, 4, 6, 24, 48, and 72 on Days 1, 29, 50, and 54 and predose on Days 8, 10, 15, 22, 33, 36, 43, and 57
Population: PK Evaluable Population. Here number of participants analyzed (N) = participants with baseline and at least 1 post baseline assessment for this outcome.
Measure: Number; unit: participants
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Number analyzed (Participants) | 7 | 13 | 9
participants
  Total GDC-0449 | 0 | 1 | 4
  Unbound GDC-0449 | 0 | 6 | 9

6. Primary Outcome: Ratio of Total and Unbound Trough GDC-0449 Concentration Between Day 57 to Day 15
Description: Ratio = trough concentration on Day 57 divided by trough concentration on Day 15. If the ratio of total and unbound trough GDC-0449 concentration between Day 57 to Day 15 is less than 1, then it indicates reduction in total and unbound trough GDC-0449 concentration between Day 15 to Day 57.
Time Frame: Predose and 1, 2, 4, 6, 24, 48, and 72 on Days 1, 29, 50, and 54 and predose on Days 8, 10, 15, 22, 33, 36, 43, and 57
Population: The PK Evaluable Population. N = participants who completed Day 57 of the study were included in this analysis.
Measure: Mean (Full Range); unit: ratio
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Number analyzed (Participants) | 7 | 13 | 9
ratio
  Css,trough for Total GDC-0449 | 1.23 [1.01 to 1.73] | 0.87 [0.49 to 1.27] | 0.54 [0.47 to 0.66]
  Css,trough for Unbound GDC-0449 | 1.34 [0.96 to 2.21] | 0.58 [0.28 to 1.49] | 0.20 [0.11 to 0.35]

7. Primary Outcome: Plasma Concentration at Steady State (Css) for Total and Unbound GDC-0449
Description: Plasma GDC-0449 concentrations were reported in nanogram per milliliter (ng/mL) units and converted to micromolar (mcM) units using the molecular weight (421.30 grams per mole [g/mol]) prior to PK analysis. Css was calculated for Days 28 to 56.
Time Frame: Predose and 1, 2, 4, 6, 24, 48, and 72 on Days 1, 29, 50, and 54 and predose on Days 8, 10, 15, 22, 33, 36, 43, and 57
Population: PK Evaluable Population. N = participants with baseline and post baseline data available for measurement of Css at steady state.
Measure: Mean (Standard Deviation); unit: mcM
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Number analyzed (Participants) | 15 | 18 | 18
mcM
  Total GDC-0449 | 28 (11.4) | 26.1 (11.8) | 16.9 (5.89)
  Unbound GDC-0449 | 0.163 (0.056) | 0.088 (0.0408) | 0.0489 (0.0259)

8. Primary Outcome: Maximum Plasma Concentration (Cmax) of Total and Unbound GDC-0449
Description: Plasma GDC-0449 concentrations were reported in ng/mL units and converted to mcM units using the molecular weight (421.30 g/mol) prior to PK analysis.
Time Frame: 0, 1, 2, 4, 6, 24, 48, 72 hours on Day 1, 15 and 57 post-dose
Population: PK Evaluable Population. 'n' signifies number of participants with data available at specified timepoint in each group.
Measure: Mean (Standard Deviation); unit: mcM
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Number analyzed (Participants) | 20 | 21 | 22
mcM
  Cmax,Total GDC-0449: Single Dose (n=20,21,22) | 7.09 (3.66) | 8.08 (3.48) | 7.29 (3.24)
  Cmax,Total GDC-0449: Day 29-36 (n=15,18,18) | 30.4 (11.6) | 29.5 (12.6) | 21.2 (5.59)
  Cmax,Total GDC-0449: Day 50-57 (n=11,13,10) | 33.9 (12.2) | 28.6 (13.8) | 18.2 (4.23)
  Cmax,Unbound GDC-0449: Single Dose (n=20,21,22) | 0.02 (0.02) | 0.02 (0.02) | 0.02 (0.01)
  Cmax,Unbound GDC-0449:Day 29-36 (n=15,18,18) | 0.215 (0.0797) | 0.122 (0.0602) | 0.0998 (0.0516)
  Cmax,Unbound GDC-0449:Day 50-57 (n=11,13,10) | 0.247 (0.0841) | 0.132 (0.0717) | 0.0688 (0.0312)

9. Primary Outcome: Area Under the Curve From Time Zero to 24 Hour (AUC0-24) for Total and Unbound GDC-0449
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. AUC values were calculated using the linear trapezoidal method when the concentrations were rising and using the logarithmic trapezoidal method when the concentrations were declining (linear up/log down rule in WinNonlin). Below the limit of quantitation (BLQ) values at pre-dose were considered as zero for PK analysis.
Time Frame: Predose and 1, 2, 4, 6, 24, 48, and 72 on Days 1, 29, 50, and 54 and predose on Days 8, 10, 15, 22, 33, 36, 43, and 57
Population: PK Evaluable Population. n = number of participants with data available at specified timepoint in each group.
Measure: Mean (Standard Deviation); unit: mcM*hour
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Number analyzed (Participants) | 20 | 21 | 22
mcM*hour
  AUC0-24,Total GDC-0449: Single Dose (n=20,21,22) | 130.88 (73.69) | 129.44 (71.66) | 126.05 (61.73)
  AUC0-24,Total GDC-0449: Day 29 (n=14,17,18) | 696 (258) | 595 (241) | 455 (116)
  AUC0-24,Total GDC-0449: Day 50 (n=11,13,9) | 729 (251) | 587 (274) | 387 (86)
  AUC0-24,Unbound GDC-0449: Single Dose (n=20,21,22) | 0.38 (0.31) | 0.30 (0.27) | 0.32 (0.20)
  AUC0-24,Unbound GDC-0449:Day 29 (n=14,17,17) | 4.06 (1.13) | 2.39 (1.29) | 1.81 (0.958)
  AUC0-24,Unbound GDC-0449:Day 50 (n=11,13,9) | 4.8 (1.75) | 2.44 (1.19) | 1.51 (0.615)

10. Primary Outcome: Area Under the Curve From Time Zero to the Last Measured Concentration (AUClast) for Total and Unbound GDC-0449
Description: AUC values were calculated using the linear trapezoidal method when the concentrations were rising and using the logarithmic trapezoidal method when the concentrations were declining (linear up/log down rule in WinNonlin). BLQ values at pre-dose were considered as zero for PK analysis.
Time Frame: Predose and 1, 2, 4, 6, 24, 48, and 72 on Days 1, 29, 50, and 54 and predose on Days 8, 10, 15, 22, 33, 36, 43, and 57
Population: PK Evaluable Population. n = number of participants with data available at specified time point in each group.
Measure: Mean (Standard Deviation); unit: mcM*hour
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Number analyzed (Participants) | 20 | 21 | 22
mcM*hour
  AUClast,Total GDC-0449: Single Dose (n=20,21,22) | 431.20 (201.18) | 478.38 (212.88) | 453.14 (209.48)
  AUClast,Total GDC-0449: Day 28-35 (n=14,14,18) | 4834.06 (1708.27) | 4302.84 (1691.87) | 2935.33 (926.74)
  AUClast,Total GDC-0449: Day 49-56 (n=9,13,9) | 5235.09 (2010.93) | 4074.88 (1779.33) | 2656.65 (666.09)
  AUClast,Unbound GDC-0449: Single Dose (n=20,21,22) | 1.19 (0.73) | 1.08 (0.82) | 1.09 (0.65)
  AUClast,Unbound GDC-0449:Day 28-35 (n=14,17,17) | 28.32 (8.37) | 15.69 (7.79) | 10.50 (6.08)
  AUClast,Unbound GDC-0449:Day 49-56 (n=8,13,9) | 33.40 (11.91) | 15.57 (6.52) | 8.76 (3.23)

11. Secondary Outcome: Duration of Response (DR)
Description: DR during first line therapy is defined as the time from when response (complete response [CR] or partial response [PR]) was first documented to first documented disease progression or death (whichever occurs first) during first line therapy. This was only be calculated for participants who achieved a best overall response of CR or PR. Participants who did not progress or die after they had a confirmed response were censored at the date of their last tumor measurement or last follow up for progression of disease during first line therapy. CR: disappearance of all target lesions (TLs) with any pathological lymph nodes (whether target or non-target) having a reduction in short axis to less than 10 millimeters. PR: at least a 30% decrease in the sum of diameters of TLs, with reference to baseline sum diameters. DR was not calculated as only 1 responding participant reached their response at the last scheduled response assessment, hence follow-up data are not available.
Time Frame: Screening Day 57, and every 8 weeks thereafter up to 52 weeks
Reporting Status: Not Posted

12. Primary Outcome: Time to Achieve Maximum Observed Plasma Concentration (Tmax) After a Single Dose of GDC-0449
Time Frame: 0, 1, 2, 4, 6, 24, 48, 72 hours on Day 1
Population: PK Evaluable Population.
Measure: Median (Full Range); unit: hours
Groups:
- GDC-0449 150 mg: All Participants: All participants received single dose of GDC-0449 150 mg capsule orally on Day 1.
Arm/Group | GDC-0449 150 mg: All Participants
Number analyzed (Participants) | 63
hours
  Total GDC-0449 | 48 [1 to 72]
  Unbound GDC-0449 | 48 [1 to 72]

ADVERSE EVENTS:
Time Frame: From signature of informed consent up to 30 days after last dose of study medication (maximum 57 days on study medication).
Description: Safety Population included all participants who received at least 1 dose of study medication.
Arm/Group | GDC-0449 150 mg QD | GDC-0449 150 mg TIW | GDC-0449 150 mg QW
Serious Adverse Events (participants affected / at risk) | 6/20 | 8/21 | 8/22
Other Adverse Events (participants affected / at risk) | 19/20 | 19/21 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GDC-0449 150 mg QD (N=20) | GDC-0449 150 mg TIW (N=21) | GDC-0449 150 mg QW (N=22)
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Jejunal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 2 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GDC-0449 150 mg QD (N=20) | GDC-0449 150 mg TIW (N=21) | GDC-0449 150 mg QW (N=22)
Nausea (Gastrointestinal disorders) | 11 | 8 | 8
Vomiting (Gastrointestinal disorders) | 7 | 3 | 8
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 6
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 5
Constipation (Gastrointestinal disorders) | 4 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 1
Ascites (Gastrointestinal disorders) | 3 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1
Faeces hard (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 8 | 8 | 9
Oedema peripheral (General disorders) | 3 | 2 | 3
Pain (General disorders) | 1 | 3 | 1
Early satiety (General disorders) | 4 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 1
Chills (General disorders) | 0 | 2 | 1
Pyrexia (General disorders) | 1 | 0 | 2
Asthenia (General disorders) | 1 | 1 | 0
Catheter site pain (General disorders) | 1 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 1
Oedema (General disorders) | 2 | 0 | 0
Suprapubic pain (General disorders) | 1 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Weight decreased (Investigations) | 4 | 4 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 5 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 4 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 3
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 1
Blood chloride decreased (Investigations) | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 3
Headache (Nervous system disorders) | 1 | 3 | 3
Dysgeusia (Nervous system disorders) | 2 | 4 | 0
Hypogeusia (Nervous system disorders) | 2 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 2
Candidiasis (Infections and infestations) | 1 | 0 | 1
Infection (Infections and infestations) | 0 | 2 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 3
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 3
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 2 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.